CLINICAL TRIAL: NCT06236178
Title: Comparing Autologous Blood, Corticosteroid, and Their Combined Injection for Treating Lateral Epicondylitis: A Randomized Clinical Trial
Brief Title: Comparing Autologous Blood, Corticosteroid, and Their Combined Injection for Treating Lateral Epicondylitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Albert ÇAKAR, MD, Orthopedic and Traumatology Surgeon, Istanbul Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: TR13734
Record Dates: First submitted 2024-01-09; First posted 2024-02-01 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Lateral Epicondylitis; Comparing Autologous Blood Corticosteroid and Their Combined Injection for Treating Lateral Epicondylitis
MeSH Terms: conditions — Tennis Elbow | interventions — Adrenal Cortex Hormones; Blood Transfusion, Autologous; Anesthetics, Local

STUDY DESIGN:
Intervention Model Description: A Randomized Clinical Trial
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Autologous Blood Injection Mixed With Local Anesthetic (Active Comparator): Autologous Blood Injection group were administered 1ml of autologous venous blood mixed with 2ml of 2% prilocaine HCl(Priloc %2,Vem,Turkey) subcutaneously.
  Interventions: Drug: Autologous Blood; Drug: Local Anesthetic
- Corticosteroid Injection Mixed With Local Anesthetic (Active Comparator): Corticosteroid Injection category were given 1ml of 40 mg methylprednisolone acetate(Prednol-L 40mg,Mustafa Nevzat,Turkey) mixed with 2ml of 2% prilocaine HCl(Priloc %2,Vem,Turkey) subcutaneously.
  Interventions: Drug: Corticosteroid; Drug: Local Anesthetic
- Combined Injection Mixed With Local Anesthetic (Active Comparator): Combined Injection group received a mixture containing 1ml each of autologous venous blood and 40mg methylprednisolone acetate(Prednol-L 40mg,Mustafa Nevzat,Turkey), along with 1ml of 2% prilocaine HCl(Priloc %2,Vem,Turkey) subcutaneously.
  Interventions: Drug: Corticosteroid; Drug: Autologous Blood; Drug: Local Anesthetic

INTERVENTIONS:
Drug: Corticosteroid — 1 ml of 40 mg methylprednisolone acetate
  Arms: Combined Injection Mixed With Local Anesthetic; Corticosteroid Injection Mixed With Local Anesthetic
Drug: Autologous Blood — 1 ml of autologous venous blood
  Arms: Autologous Blood Injection Mixed With Local Anesthetic; Combined Injection Mixed With Local Anesthetic
Drug: Local Anesthetic — 1 ml of 2% prilocaine HCl

SUMMARY:
The goal of this clinical trial is to compare autologous blood, corticosteroid, and their combined injection for treating lateral epicondylitis. The main question it aims to answer are:

• Which of these highly used drugs in treatment of lateral epicondylitis is more effective? Participants were randomly allocated into three equal treatment groups (AB versus CS versus their combination) with sealed envelopes prepared by a computer-based random number generator. Patients in the AB Group received 1 ml of autologous venous blood mixed with 2 ml of 2% prilocaine HCl, patients in the CS Group received 1 ml of 40 mg methylprednisolone acetate mixed with 2 ml of 2% prilocaine HCl, and patients in the Combined Group (AB+CS) received 1 ml of autologous venous blood, 1 ml of 40 mg methylprednisolone acetate mixed with 1 ml of 2% prilocaine HCl. Each group received an equal amount of (3 ml) injected material. PRTEE and HGS measurements were assessed before the injection (baseline values), on Day 15, Day 30, and Day 90, in the same manner by the senior author.

DETAILED DESCRIPTION:
This study aimed to compare the efficacy of autologous blood (AB) and corticosteroid (CS) injections and their combination in treating lateral epicondylitis (LE), hypothesizing that the combined approach might offer immediate symptom resolution and lower recurrence. Methods: A total of 120 patients diagnosed with lateral epicondylitis were systematically distributed among three distinct therapeutic injection groups. Those in the AB group were administered 1ml of autologous venous blood mixed with 2ml of 2% prilocaine HCl. Participants in the CS category were given 1ml of 40 mg methylprednisolone acetate mixed with 2ml of 2% prilocaine HCl. Meanwhile, patients in the combined group received a mixture containing 1ml each of autologous venous blood and 40mg methylprednisolone acetate, along with 1ml of 2% prilocaine HCl. Prior to receiving their respective injections, a comprehensive assessment of all participants was carried out. Follow-up assessments were subsequently conducted on days 15, 30, and 90, utilizing metrics of patient-rated tennis elbow evaluation (PRTEE) and measurements of hand grip strength (HGS).

ELIGIBILITY:
Inclusion Criteria:

1-Patients with LE whose complaints persisted for more than 3 months

Exclusion Criteria:

1. Patients with a history of recent trauma,
2. Congenital or neuromuscular disease or abnormality of the upper limb
3. Previous upper limb surgery,
4. History of rheumatic disease,
5. History of cervical disc pathology or carpal tunnel syndrome
6. Systemic corticosteroid treatment
7. Any previous local injection treatment
8. Patients with a history of previous allergic reaction towards local anesthetics and corticosteroids

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 119 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Patient-rated tennis elbow evaluation questionnaire (PRTEE) scores | Before the injection (baseline values), on Day 15, Day 30, and Day 90
  Patient-rated tennis elbow evaluation questionnaire (PRTEE) is consist of 2 steps, pain and function score.
  Pain Score is measured by sum of the 5 pain items (out of 50) (Best Score = 0, Worst Score = 50) Function Score is measured by sum of the of the 10 function items, divided by 2 (out of 50) (Best Score = 0, Worst Score = 50) Total Score is measured by sum of pain and function scores(Best Score = 0, Worst Score = 100)

SECONDARY OUTCOMES:
Hand Grip Strength (HGS) measurements | Before the injection (baseline values), on Day 15, Day 30, and Day 90
  Hand grip strength (HGS) was measured with a digital hand dynamometer before and on Day 15, Day 30, and Day 90 after injection in all patients.

CONTACTS AND LOCATIONS:
Overall Officials: Albert ÇAKAR, MD, Principal Investigator — Istanbul Training and Research Hospital
Locations (2):
- Turkey (Türkiye) (2):
  - Istanbul Training and Research Hospital, Department of Orthopedics and Traumatology,, Istanbul
  - Istanbul Training and Research Hospital, Istanbul

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: SAP

REFERENCES:
- [Background] Defoort S, De Smet L, Brys P, Peers K, Degreef I. Lateral elbow tendinopathy: surgery versus extracorporeal shock wave therapy. Hand Surg Rehabil. 2021 Jun;40(3):263-267. doi: 10.1016/j.hansur.2020.12.008. Epub 2021 Feb 23. PMID 33636381
- [Background] Nirschl RP. Elbow tendinosis/tennis elbow. Clin Sports Med. 1992 Oct;11(4):851-70. PMID 1423702
- [Background] Krogh TP, Bartels EM, Ellingsen T, Stengaard-Pedersen K, Buchbinder R, Fredberg U, Bliddal H, Christensen R. Comparative effectiveness of injection therapies in lateral epicondylitis: a systematic review and network meta-analysis of randomized controlled trials. Am J Sports Med. 2013 Jun;41(6):1435-46. doi: 10.1177/0363546512458237. Epub 2012 Sep 12. PMID 22972856
- [Background] Kivrak A, Ulusoy I. Comparison of the Clinical Results of Platelet-Rich Plasma, Steroid and Autologous Blood Injections in the Treatment of Chronic Lateral Epicondylitis. Healthcare (Basel). 2023 Mar 6;11(5):767. doi: 10.3390/healthcare11050767. PMID 36900772
- [Background] Goorens CK, Wernaers P, Dewaele J. Standardized Tendon Fenestration with Injection of Autologous Blood for Treatment of Lateral Epicondylitis. J Hand Microsurg. 2020 Sep 17;14(3):240-244. doi: 10.1055/s-0040-1716991. eCollection 2022 Jul. PMID 36016641
- [Background] Tang S, Wang X, Wu P, Wu P, Yang J, Du Z, Liu S, Wei F. Platelet-Rich Plasma Vs Autologous Blood Vs Corticosteroid Injections in the Treatment of Lateral Epicondylitis: A Systematic Review, Pairwise and Network Meta-Analysis of Randomized Controlled Trials. PM R. 2020 Apr;12(4):397-409. doi: 10.1002/pmrj.12287. Epub 2020 Jan 13. PMID 31736257
- [Background] Arirachakaran A, Sukthuayat A, Sisayanarane T, Laoratanavoraphong S, Kanchanatawan W, Kongtharvonskul J. Platelet-rich plasma versus autologous blood versus steroid injection in lateral epicondylitis: systematic review and network meta-analysis. J Orthop Traumatol. 2016 Jun;17(2):101-12. doi: 10.1007/s10195-015-0376-5. Epub 2015 Sep 11. PMID 26362783
- [Background] Kinney WR, Anderson BR. Nonoperative Management of Lateral Epicondyle Tendinopathy: An Umbrella Review. J Chiropr Med. 2023 Sep;22(3):204-211. doi: 10.1016/j.jcm.2023.04.004. Epub 2023 Jul 10. PMID 37644995
- [Background] Edwards SG, Calandruccio JH. Autologous blood injections for refractory lateral epicondylitis. J Hand Surg Am. 2003 Mar;28(2):272-8. doi: 10.1053/jhsu.2003.50041. PMID 12671860
- [Background] Kazemi M, Azma K, Tavana B, Rezaiee Moghaddam F, Panahi A. Autologous blood versus corticosteroid local injection in the short-term treatment of lateral elbow tendinopathy: a randomized clinical trial of efficacy. Am J Phys Med Rehabil. 2010 Aug;89(8):660-7. doi: 10.1097/PHM.0b013e3181ddcb31. PMID 20463564
- [Background] Ozturan KE, Yucel I, Cakici H, Guven M, Sungur I. Autologous blood and corticosteroid injection and extracoporeal shock wave therapy in the treatment of lateral epicondylitis. Orthopedics. 2010 Feb;33(2):84-91. doi: 10.3928/01477447-20100104-09. PMID 20192142
- [Background] MacDermid JC, Turgeon T, Richards RS, Beadle M, Roth JH. Patient rating of wrist pain and disability: a reliable and valid measurement tool. J Orthop Trauma. 1998 Nov-Dec;12(8):577-86. doi: 10.1097/00005131-199811000-00009. PMID 9840793
- [Background] Altan L, Ercan I, Konur S. Reliability and validity of Turkish version of the patient rated tennis elbow evaluation. Rheumatol Int. 2010 Jun;30(8):1049-54. doi: 10.1007/s00296-009-1101-6. Epub 2009 Aug 26. PMID 19707766
- [Background] Poltawski L, Watson T. Measuring clinically important change with the Patient-rated Tennis Elbow Evaluation. Hand Therapy. 2011;16(3):52-57. https://doi.org/ 10.1258/ht.2011.011013
- [Background] Fess EE. Grip strength. In: Casanova JS, editor. Clinical assessment recommendations, Chicago: American Society of Hand Therapists;1992; p. 41-5.
- [Background] BAILY RA, BROCK BH. Hydrocortisone in tennis elbow; a controlled series. Proc R Soc Med. 1957 Jun;50(6):389-90. doi: 10.1177/003591575705000605. No abstract available. PMID 13453415
- [Background] Judson CH, Wolf JM. Lateral epicondylitis: review of injection therapies. Orthop Clin North Am. 2013 Oct;44(4):615-23. doi: 10.1016/j.ocl.2013.06.013. Epub 2013 Aug 21. PMID 24095076
- [Background] Wolf JM, Ozer K, Scott F, Gordon MJ, Williams AE. Comparison of autologous blood, corticosteroid, and saline injection in the treatment of lateral epicondylitis: a prospective, randomized, controlled multicenter study. J Hand Surg Am. 2011 Aug;36(8):1269-72. doi: 10.1016/j.jhsa.2011.05.014. Epub 2011 Jun 25. PMID 21705157
- [Background] Dojode CM. A randomised control trial to evaluate the efficacy of autologous blood injection versus local corticosteroid injection for treatment of lateral epicondylitis. Bone Joint Res. 2012 Aug 1;1(8):192-7. doi: 10.1302/2046-3758.18.2000095. Print 2012 Aug. PMID 23610690
- [Background] Jindal N, Gaury Y, Banshiwal RC, Lamoria R, Bachhal V. Comparison of short term results of single injection of autologous blood and steroid injection in tennis elbow: a prospective study. J Orthop Surg Res. 2013 Apr 27;8:10. doi: 10.1186/1749-799X-8-10. PMID 23621906
- [Background] Arik HO, Kose O, Guler F, Deniz G, Egerci OF, Ucar M. Injection of autologous blood versus corticosteroid for lateral epicondylitis: a randomised controlled study. J Orthop Surg (Hong Kong). 2014 Dec;22(3):333-7. doi: 10.1177/230949901402200313. PMID 25550013
- [Background] Branson R, Naidu K, du Toit C, Rotstein AH, Kiss R, McMillan D, Fooks L, Coombes BK, Vicenzino B. Comparison of corticosteroid, autologous blood or sclerosant injections for chronic tennis elbow. J Sci Med Sport. 2017 Jun;20(6):528-533. doi: 10.1016/j.jsams.2016.10.010. Epub 2016 Oct 29. PMID 28089102
- [Background] Kaya SS, Yardimci G, Goksu H, Genc H. Effects of splinting and three injection therapies (corticosteroid, autologous blood and prolotherapy) on pain, grip strength, and functionality in patients with lateral epicondylitis. Turk J Phys Med Rehabil. 2022 Jun 1;68(2):205-213. doi: 10.5606/tftrd.2022.8007. eCollection 2022 Jun. PMID 35989952
- [Background] Lee SH, Choi HH, Chang MC. The effects of inclusion of minimal-dose corticosteroid in autologous whole blood and dextrose injection for the treatment of lateral epicondylitis. J Back Musculoskelet Rehabil. 2022;35(1):129-134. doi: 10.3233/BMR-200261. PMID 34151824
- [Derived] Cakar A, Gozlu OD. Comparing autologous blood, corticosteroid, and a combined injection of both for treating lateral epicondylitis: a randomized clinical trial. J Orthop Traumatol. 2024 Jul 4;25(1):34. doi: 10.1186/s10195-024-00772-4. PMID 38963583

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-01-19): https://cdn.clinicaltrials.gov/large-docs/78/NCT06236178/Prot_SAP_000.pdf
  • Informed Consent Form (2024-01-29): https://cdn.clinicaltrials.gov/large-docs/78/NCT06236178/ICF_001.pdf